CLINICAL TRIAL: NCT03522389
Title: The Effect of Action Observation Training on Gait Variables and Global Cognitive Functions in Older Adult With Mild Cognitive Impairment: A Randomized Controlled Trial
Brief Title: Effect of Action Observation Training on Gait Variables and Global Cognitive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MU-CIRB 2018/001.0301
Record Dates: First submitted 2018-04-17; First posted 2018-05-11 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Action Observation Training; Gait
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AOT with gait training group (Experimental): Action observation training with gait training
  Interventions: Procedure: AOT with gait training
- Gait training group (Active Comparator): Gait training
  Interventions: Procedure: Gait training
- Control group (Other): Education
  Interventions: Other: Education

INTERVENTIONS:
Procedure: AOT with gait training — AOT with gait training composes of program of watching video in different views of normal walk for 5 min.
  After that, participants will receive gait training program. The program consists of warm-up, gait training, cool-down, and stretching. Gait training is classified into the different levels of difficulty in each week. The 1st week will be walking over the markers followed by 100 steps/min of metronome. The second week will be walking over the markers followed by 120 step/min of metronome. The 3rd week will be walking followed by 120 step/min of metronome but not has the markers. The 4th week will imagine and imitate the walking in the 2nd week but not has the markers and metronome.
  Arms: AOT with gait training group
Procedure: Gait training — To control a total time of training, the gait training group will watch video of Vincent van Gogh's painting for 5 min. After that, participants will training the gait as protocol of experimental group.
  The program consists of warm-up, gait training, cool-down, and stretching. Gait training is classified into the different levels of difficulty in each week. The 1st week will be walking over the markers followed by 100 steps/min of metronome. The second week will be walking over the markers followed by 120 step/min of metronome. The 3rd week will be walking followed by 120 step/min of metronome but not has the markers. The 4th week will imagine and imitate the walking in the 2nd week but not has the markers and metronome.
  Arms: Gait training group
Other: Education — There will be no intervention exercise program provide for the control group. They will receive education about dementia such as definition, etiology, sign and symptom, and caring.
  Arms: Control group

SUMMARY:
This study will investigate the effect of Action Observation Teaining (AOT) on gait variables and global cognitive functions in older adults with mild cognitive impairment (MCI).

The specific objectives are 1) to compare gait variables and global cognitive functions among the AOT with gait training, gait training, and control groups at before training, after training, and follow up and 2) to compare gait variables and global cognitive functions among before training, after training, and follow up in each of the groups.

DETAILED DESCRIPTION:
Participants in this study will be older adults recruiting from the Physical Therapy Center of Mahidol University, Siriraj hospital, and community at Phuttamonthon area (n = 39).

They will be diagnosed as a MCI, using core clinical criteria of the National Institute on Aging and the Alzheimer's Association by a physiotherapist. Prior to participate in the study, participants will be informed the details of the study and sign the informed consent. All participants will be recorded the demographic data and will be assessed visual acuity, hearing, sensation and muscle strength of lower extremity, balance, gait variables, and global cognitive function.

Participants who pass the criteria will be randomly assigned to either the AOT with gait training group (n = 13), the gait training group (n = 13), and the control group (n = 13) by stratified randomization.

Gait variables will be collected by the Force Distribution Measurement platform during walking at comfortable speed (single task) and during counting backwards from 100 by sevens (dual tasks). Global cognitive function will be assessed by the Montral Cognitve Assessment (MoCA).

All varaibles will be assessed 3 times which will be at before training, after 4-week of training, and 4-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60-80 years old.
* Having subjective evidence of cognitive decline from patients, or from closely informants, or from a clinicians.
* Having objective evidence of cognitive decline, deﬁned by using a Montreal Cognitive Assessment (MoCA) 18-24 points.
* Independent function in daily life
* Independent walking without using gait aids.
* Having fall risk, defined by the fall risk threshold (gait velocity < 1 m/s in walking while counting backwards from 100 by sevens).
* Able to understand Thai language and follow study protocol.

Exclusion Criteria:

* Having history of stroke or heart attack or Parkinsonism symptoms.
* The presence of major depression disorder deﬁned by a Patient Health Questionnaire-9 > 9 points.
* Diagnosis as dementia by neurologists.
* Any cardiac or respiratory disease that could cause gait limiting.
* Musculoskeletal disorder that affected gait performance.
* Balance disorder in assessment day, such as vertigo and dizziness.
* Visual acuity with a glasses worse than 6/15 (metric system) in both their eyes.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rommanee Rojasavastera, Principal Investigator — Faculty of Physical Therapy, Mahidol University
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montero-Odasso M, Muir SW, Speechley M. Dual-task complexity affects gait in people with mild cognitive impairment: The interplay between gait variability, dual tasking, and risk of falls. Arch Phys Med Rehabil. 2012;93(2):293-9. Park H, Kim J, Lee M, Oh D. Clinical feasibility of action observation training for walking function of patients with post-stroke hemiparesis: a randomized controlled trial. Clin Rehabil. 2014;28(8):794-803. Scherder E, Eggermont L, Visscher C, Scheltens P, Swaab D. Understanding higher level gait disturbances in mild dementia in order to improve rehabilitation: 'Last in-first out'. Neurosci Biobehav Rev. 2011;35(3):699-714. Beauchet O, Launay CP, Annweiler C, Allali G. Hippocampal volume, early cognitive decline and gait variability: Which association? Exp Gerontol. 2015;61:98-104.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 97 participants initially assessed for eligibility, 58 were excluded: 55 did not meet the inclusion criteria and 3 declined to participate. Therefore, 39 participants were enrolled and randomly assigned to one of the three groups.
Groups:
- AOT With Gait Training Group: Action observation training with gait training
  AOT with gait training: AOT with gait training composes of program of watching video in different views of normal walk for 5 min.
  After that, participants will receive gait training program. The program consists of warm-up, gait training, cool-down, and stretching. Gait training is classified into the different levels of difficulty in each week. The 1st week will be walking over the markers followed by 100 steps/min of metronome. The second week will be walking over the markers followed by 120 step/min of metronome. The 3rd week will be walking followed by 120 step/min of metronome but not has the markers. The 4th week will imagine and imitate the walking in the 2nd week but not has the markers and metronome.
- Gait Training Group: Gait training
  Gait training: To control a total time of training, the gait training group will watch video of Vincent van Gogh's painting for 5 min. After that, participants will training the gait as protocol of experimental group.
  The program consists of warm-up, gait training, cool-down, and stretching. Gait training is classified into the different levels of difficulty in each week. The 1st week will be walking over the markers followed by 100 steps/min of metronome. The second week will be walking over the markers followed by 120 step/min of metronome. The 3rd week will be walking followed by 120 step/min of metronome but not has the markers. The 4th week will imagine and imitate the walking in the 2nd week but not has the markers and metronome.
Period: Overall Study
Arm/Group | AOT With Gait Training Group | Gait Training Group | Control Group
Started | 13 | 13 | 13
Completed | 11 | 11 | 11
Not Completed | 2 | 2 | 2
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — had herniated nucleus pulposus | 0 | 1 | 0
Not completed — go to work in other province | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AOT With Gait Training Group | Gait Training Group | Control Group | Total
Number analyzed (Participants) | 11 | 11 | 11 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.64 (4.64) | 67.50 (5.60) | 65.71 (2.45) | 66.92 (4.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 8 | 25
  Male | 2 | 3 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.08 (3.19) | 24.71 (3.69) | 25.38 (3.80) | 24.72 (3.57)

OUTCOME MEASURES:

1. Primary Outcome: Gait Speed During the Single Task
Description: Gait speed during the single-task condition was measured in meter per second while participants walked at a comfortable pace over a measurement platform without performing any secondary task. Higher gait speed values indicate better physical function and mobility, whereas lower values may reflect impaired motor performance or increased risk of functional decline.
  Unit of Measure: meters per second (m/s)
Time Frame: Baseline (T1), After 4 weeks of training (T2), and 1-month follow-up (T3)
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | AOT With Gait Training Group | Gait Training Group | Control Group
Number analyzed (Participants) | 11 | 11 | 11
m/s
  After 4 weeks of training - Baseline (T2-T1) | 0.17 (0.10) | 0.09 (0.12) | 0.00 (0.08)
  1-month follow-up - Baseline (T3-T1) | 0.15 (0.09) | 0.12 (0.08) | -0.01 (0.10)
  Baseline (T1) | 0.86 (0.16) | 0.94 (0.14) | 0.88 (0.15)
  After 4 weeks of training (T2) | 1.02 (0.15) | 1.03 (0.10) | 0.88 (0.15)
  1-month follow-up (T3) | 1.01 (0.15) | 1.06 (0.10) | 0.87 (0.17)
Statistical Analysis 1: Comparison: AOT With Gait Training Group vs Gait Training Group vs Control Group; After 4 weeks of training - Baseline (T2-T1); Test type: Superiority; p = 0.003, ANOVA
Statistical Analysis 2: Comparison: AOT With Gait Training Group vs Gait Training Group vs Control Group; 1-month follow up - Baseline (T3-T1); Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: AOT With Gait Training Group; Within group comparison; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 4: Comparison: Gait Training Group; Within group comparison; Test type: Superiority; p = 0.006, ANOVA
Statistical Analysis 5: Comparison: Control Group; Within group comparison; Test type: Superiority; p = 0.793, ANOVA

2. Primary Outcome: Gait Speed During the Dual Task
Description: Gait speed during the dual-task condition was measured in meters per second (m/s), while participants walked at a comfortable pace over a measurement platform while simultaneously counting a number backward by 7. Higher gait speed values indicate better cognitive-motor performance, while lower values suggest impaired dual-task ability and potential functional or cognitive decline.
  Unit of Measure: meters per second (m/s).
Time Frame: Baseline (T1), After 4 weeks of training (T2), and 1-month follow-up (T3)
Measure: Mean (Standard Error); unit: m/s
Arm/Group | AOT With Gait Training Group | Gait Training Group | Control Group
Number analyzed (Participants) | 11 | 11 | 11
m/s
  After 4 weeks of training - Baseline (T2-T1) | 0.17 (0.07) | 0.12 (0.13) | -0.02 (0.07)
  1-month follow-up - Baseline (T3-T1) | 0.15 (0.08) | 0.12 (0.13) | 0.04 (0.10)
  Baseline (T1) | 0.69 (0.17) | 0.70 (0.24) | 0.64 (0.18)
  After 4 weeks of training (T2) | 0.86 (0.22) | 0.82 (0.24) | 0.62 (0.19)
  1-month follow-up (T3) | 0.84 (0.23) | 0.82 (0.23) | 0.68 (0.18)
Statistical Analysis 1: Comparison: AOT With Gait Training Group vs Gait Training Group vs Control Group; After 4 weeks of training - Baseline (T2-T1); Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: AOT With Gait Training Group vs Gait Training Group vs Control Group; 1-month follow-up - Baseline (T3-T1); Test type: Superiority; p = 0.039, ANOVA
Statistical Analysis 3: Comparison: AOT With Gait Training Group; Within group comparison; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 4: Comparison: Gait Training Group; Within group comparison; Test type: Superiority; p = 0.002, ANOVA
Statistical Analysis 5: Comparison: Control Group; Within group comparison; Test type: Superiority; p = 0.117, ANOVA

3. Secondary Outcome: Stride Time Variability During Single Task
Description: Stride time variability during single task was measured while participants walked at a comfortable pace over a measurement platform. Stride time refers to the duration between successive heel contacts of the same foot. The variability of stride time was quantified using the coefficient of variation (CV), calculated as: (standard deviation of stride time / mean stride time) × 100. Higher CV values indicate greater variability in stride timing, which reflects reduced gait stability or impaired coordination. Lower CV values are considered better outcomes, indicating more stable and consistent gait.
  Unit of Measure: percentage of coefficient of variation (% Cov).
Time Frame: Baseline (T1), After 4 weeks of training (T2), and 1-month follow-up (T3)
Measure: Mean (Standard Deviation); unit: %Cov
Arm/Group | AOT With Gait Training Group | Gait Training Group | Control Group
Number analyzed (Participants) | 11 | 11 | 11
%Cov
  After 4 weeks of training - Baseline (T2-T1) | 0.06 (1.49) | 0.01 (0.89) | 0.20 (0.95)
  1-month follow-up - Baseline (T3-T1) | -0.09 (1.73) | -0.05 (1.19) | -0.34 (0.69)
  Baseline (T1) | 2.42 (1.15) | 1.85 (0.78) | 2.67 (0.98)
  After 4 weeks of training (T2) | 2.48 (0.73) | 1.86 (0.71) | 2.87 (1.21)
  1-month follow-up (T3) | 2.33 (0.89) | 1.80 (0.72) | 2.33 (1.12)
Statistical Analysis 1: Comparison: AOT With Gait Training Group vs Gait Training Group vs Control Group; After 4 weeks of training - Baseline (T2-T1); Test type: Superiority; p = 0.924, ANOVA
Statistical Analysis 2: Comparison: AOT With Gait Training Group vs Gait Training Group vs Control Group; 1-month follow-up - Baseline (T3-T1); Test type: Superiority; p = 0.855, ANOVA
Statistical Analysis 3: Comparison: AOT With Gait Training Group; Within group comparison; Test type: Superiority; p = 0.937, ANOVA
Statistical Analysis 4: Comparison: Gait Training Group; Within group comparison; Test type: Superiority; p = 0.970, ANOVA
Statistical Analysis 5: Comparison: Control Group; Within group comparison; Test type: Superiority; p = 0.242, ANOVA

4. Secondary Outcome: Stride Time Variability During Dual Task
Description: Stride time variability during dual-task walking was measured while participants walked at a comfortable pace, together with counting a number backward by 7 over a measurement platform. Stride time refers to the duration between successive heel contacts of the same foot. The variability of stride time was quantified using the coefficient of variation (CV), calculated as: (standard deviation of stride time / mean stride time) × 100. Higher CV values indicate greater variability in stride timing, which reflects reduced gait stability or impaired motor-cognitive coordination. Lower CV values are considered better outcomes, indicating more stable and consistent gait.
  Unit of Measure: percentage of coefficient of variation (% Cov).
Time Frame: Baseline (T1), After 4 weeks of training (T2), and 1-month follow-up (T3)
Measure: Mean (Standard Deviation); unit: % Cov
Arm/Group | AOT With Gait Training Group | Gait Training Group | Control Group
Number analyzed (Participants) | 11 | 11 | 11
% Cov
  After 4 weeks of training - Baseline (T2-T1) | -1.41 (2.50) | -0.38 (2.63) | 0.93 (3.18)
  1-month follow-up - Baseline (T3-T1) | -1.57 (2.76) | -1.15 (1.90) | 1.20 (3.55)
  Baseline (T1) | 5.30 (3.90) | 5.34 (4.93) | 5.41 (2.63)
  After 4 weeks of training (T2) | 3.89 (2.29) | 4.95 (5.95) | 6.34 (4.40)
  1-month follow-up (T3) | 3.73 (2.06) | 4.19 (4.85) | 6.61 (3.74)
Statistical Analysis 1: Comparison: AOT With Gait Training Group vs Gait Training Group vs Control Group; After 4 weeks of training - Baseline (T2-T1); Test type: Superiority; p = 0.161, ANOVA
Statistical Analysis 2: Comparison: AOT With Gait Training Group vs Gait Training Group vs Control Group; 1-month follow-up - Baseline (T3-T1); Test type: Superiority; p = 0.161, ANOVA
Statistical Analysis 3: Comparison: AOT With Gait Training Group; Within group comparison; Test type: Superiority; p = 0.076, ANOVA
Statistical Analysis 4: Comparison: Gait Training Group; Within group comparison; Test type: Superiority; p = 0.211, ANOVA
Statistical Analysis 5: Comparison: Control Group; Within group comparison; Test type: Superiority; p = 0.573, ANOVA

5. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: The Montreal Cognitive Assessment (MoCA) is a global cognitive screening tool designed to assess multiple cognitive domains, including attention, memory, language, visuospatial skills, executive function, and orientation. The test consists of 30 points in total and ranges from 0 to 30, with higher scores indicating better cognitive function.
  Unit of Measure: scores.
Time Frame: Baseline (T1), After 4 weeks of training (T2), and 1-month follow-up (T3)
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | AOT With Gait Training Group | Gait Training Group | Control Group
Number analyzed (Participants) | 11 | 11 | 11
scores
  After 4 weeks of training - Baseline (T2-T1) | 2.45 (1.63) | 1.36 (2.69) | 2.27 (1.90)
  1-month follow-up - Baseline (T3-T1) | 4.64 (1.86) | 2.36 (2.80) | 2.36 (2.29)
  Baseline (T1) | 22.18 (1.47) | 22.64 (1.36) | 22.18 (1.94)
  After 4 weeks of training (T2) | 24.64 (2.34) | 24.00 (2.86) | 24.45 (2.91)
  1-month follow-up (T3) | 26.82 (2.04) | 25.00 (3.16) | 24.54 (2.91)
Statistical Analysis 1: Comparison: AOT With Gait Training Group vs Gait Training Group vs Control Group; After 4 weeks of training - Baseline (T2-T1); Test type: Superiority; p = 0.445, ANOVA
Statistical Analysis 2: Comparison: AOT With Gait Training Group vs Gait Training Group vs Control Group; 1-month follow-up - Baseline (T3-T1); Test type: Superiority; p = 0.046, ANOVA
Statistical Analysis 3: Comparison: AOT With Gait Training Group; Within group comparison; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 4: Comparison: Gait Training Group; Within group comparison; Test type: Superiority; p = 0.028, ANOVA
Statistical Analysis 5: Comparison: Control Group; Within group comparison; Test type: Superiority; p = 0.002, ANOVA

ADVERSE EVENTS:
Time Frame: 2 months (4 weeks of intervention plus 1 month follow-up)
Arm/Group | AOT With Gait Training Group | Gait Training Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT03522389/Prot_SAP_000.pdf